CLINICAL TRIAL: NCT06544291
Title: Combination of THC and CBD as Novel Treatment for Co-Occurring Opioid Use Disorder and Chronic Pain
Brief Title: Combined THC and CBD for OUD and Chronic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Joao De Aquino, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000038372; 1R01DA060066-01 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Opioid Use Disorder
Keywords: Delta-9-Tetrahydrocannabinol; Cannabidiol; Cannabinoid; Methadone; Opioid Addiction; Pain
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This phase 2 study will utilize a double-blind, placebo-controlled, crossover experimental design. We will enroll 147 participants with co-occurring OUD and chronic pain who are receiving methadone maintenance treatment and randomize them into three groups (n=49). Across three test sessions, each group will receive single doses of THC (5 mg, 10 mg, or placebo) and CBD (300 mg, 600 mg, or placebo) in a 3x3 design, with THC dose as a between-subject (parallel-group) factor and CBD dose as within-subject (crossover) factor.
Who Masked: Participant, Investigator
Masking Description: The study medication will be prepared by the CMHC research pharmacy using over-encapsulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dronabinol 5mg (Active Comparator): Participants will be randomized to which dronabinol (or placebo) dose they receive. The fixed dose they receive will be administered across all three test sessions. Therefore, participants may receive a single capsule of 5 mg Dronabinol across all three test sessions
  Interventions: Drug: CBD 300mg; Drug: CBD 600mg; Drug: Placebo 0mg
- Dronabinol 10mg (Active Comparator): Participants will be randomized to which dronabinol (or placebo) dose they receive. The fixed dose they receive will be administered across all three test sessions. Therefore, participants may receive a single capsule of 10 mg Dronabinol across all three test sessions
  Interventions: Drug: CBD 300mg; Drug: CBD 600mg; Drug: Placebo 0mg
- Placebo 0mg (Placebo Comparator): Participants will be randomized to which dronabinol (or placebo) dose they receive. The fixed dose they receive will be administered across all three test sessions. Therefore, participants may receive a single capsule of 0 mg Dronabinol across all three test sessions
  Interventions: Drug: CBD 300mg; Drug: CBD 600mg; Drug: Placebo 0mg

INTERVENTIONS:
Drug: CBD 300mg — 3 Nantheia™ (100mg) softgel capsules and 3 placebo (0mg) softgel capsules will be administered to participants on one of the three test session days.
  Other Names: Nantheia™ ATL5 (300mg)
Drug: CBD 600mg — 6 Nantheia™ (100mg) softgel capsules will be administered to participants on one of the three test session days.
  Other Names: Nantheia™ ATL5 (600mg)
Drug: Placebo 0mg — 6 placebo (0 mg) softgel capsules will be administered to participants on one of the three test session days.
  Other Names: Nantheia™ ATL5 (0mg)

SUMMARY:
The primary objective of this phase 2 study is to investigate the therapeutic potential of orally administered combined delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) in relieving both pain and cue-induced opioid craving in people with co-occurring opioid use disorder (OUD) and chronic pain who are undergoing methadone therapy.

DETAILED DESCRIPTION:
This phase 2 study will utilize a rigorous double-blind, placebo-controlled, crossover experimental design. We will enroll 147 participants with co-occurring OUD and chronic pain who are receiving methadone maintenance treatment and randomize them into three groups (n=49). Across three test sessions, each group will receive single doses of THC (5 mg, 10 mg, or placebo) and CBD (300 mg, 600 mg, or placebo) in a 3x3 design, with THC dose as a between-subject (parallel-group) factor and CBD dose as within-subject (crossover) factor. All three groups will undergo otherwise identical procedures to ensure internal validity.

Our central hypothesis posits that, combined, THC and CBD will be more effective in alleviating pain and cue-induced opioid craving than either drug alone. While THC's analgesic effects may benefit those with co-occurring OUD and chronic pain, its abuse potential and cognitive/psychomotor deficits require careful dose consideration. Combining THC with non-hedonic and neuroprotective CBD could offer a compelling two-pronged approach to alleviate both pain and opioid craving. This study will also explore if sex influences the responses to THC and CBD, given the growing evidence indicating sex-specific effects of cannabinoids and pain responses. If our hypothesis is confirmed, selected THC/CBD doses may serve as a novel, dual-action therapy to alleviate both pain and opioid craving in co-occurring OUD and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female aged 18-65 years.
4. Co-occurring OUD (meeting DSM-5 criteria) and chronic pain (uniformly operationalized as high-impact [occurring most days, limiting life or work activities] non-cancer low back pain for ≥ 3 months).
5. Prior exposure to cannabis or its constituent cannabinoids at least once in the last 10 years, 1-10 times in the last 20 years, or more than 20 times in lifetime.
6. Adherence to their clinically prescribed methadone therapy, on a stable dose (30-150 mg/day ≥ 3 weeks).
7. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 2 weeks after the last test session.
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

1. Meeting DSM-5 criteria for cannabis use disorder and/or substance use disorders (SUDs) within the last 3 months. Participants meeting DSM-5 criteria for OUD and/or tobacco use disorder, either currently or within the last 3 months, will not be excluded per this criterion.
2. Clinically significant medical disorders as noted by the participant or through study screening procedures (e.g. liver dysfunction, as indicated by ALT and/or AST > 1.5 times the normal limit).
3. Neurological conditions that may change the response to nociceptive stimuli (e.g., stroke, neuropathy), or that lead to loss of balance, evidenced by a neuro-sensory exam during screening.
4. Contraindications for exposure to nociceptive stimuli, such as untreated hypertension, verbally noted by participant or verified during screening procedures.
5. Abnormal screening EKG (QTc interval >450 ms), arrythmia, or vasospastic disease.
6. Positive urine pregnancy test, or lack of birth control measures in women of childbearing potential. For males of reproductive potential refusal to use condoms or other methods to ensure effective contraception with partner.
7. Currently lactating.
8. Male participants who plan to donate sperm starting at screening and through 90 days after final study drug administration.
9. Females who plan to donate ova starting at screening through 28 days after final study drug administration.
10. History of primary psychotic disorders or mood disorders with psychotic features.
11. Current suicidal ideation or related behavior.
12. A physician will carefully evaluate participants for use of over-the-counter or prescription psychoactive drugs known to affect pain threshold or pain tolerance (including NSAIDS, serotonin-norepinephrine reuptake inhibitors (SNRIs) (e.g. venlafaxine, duloxetine), gabapentinoids, tricyclic antidepressants (e.g., nortriptyline, amitriptyline), anticonvulsant medications (e.g., topiramate, carbamazepine). Only participants who are on stable doses (i.e., consistent daily administration of the medication for at least three months at the same dose following the last dose change, either increase or decrease) of these medications, and whose dosing schedules allow participation in the study visits, thus excluding instances of single-dose or temporary dosing of the medication, will be eligible as determined by the sponsor-investigator. If possible, the morning dose will be administered after the study visit.
13. Current, regular use of benzodiazepines, other prescription opioids, or platelet inhibitors (e.g., clopidogrel, apixaban, ticagrelor).
14. Allergy or serious adverse reaction to cannabis or its constituent cannabinoid.
15. Allergy or serious adverse reaction to sesame oil or seeds.
16. Allergy or serious adverse reaction to Butylated Hydroxytoluene (BHT).
17. Unable to swallow or have difficulty swallowing capsules.
18. Prior to receiving the study medication on the first test session, participants' cannabinoid use will be assessed using a quantitative point-of-care urine 11-nor-9-carboxy-THC concentration test with a cut-off of ≤ 150 mg/mL. If a participant tests greater than ≤ 150 mg/mL, they will be asked to abstain for an additional 7 to 14 days. If 14 days after their initial THC concentration test the participant continues to test positive, they will not be allowed to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2028-01-28 (Estimated); Study Completion 2028-01-28 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Variable #1: Pain Sensitivity | Up to 8 hours
  We will measure pain sensitivity using a comprehensive QST battery at baseline and approximately hourly for 8 hours. The battery includes several nociceptive modalities such as pressure, mechanical, heat, and cold stimuli. The main outcome will be a composite pain sensitivity measure, integrating data from the QST battery.
Primary Outcome Variable #2: Opioid Craving | Baseline and +180 minutes post dose
  We will measure opioid craving using the short form Heroin Craving Questionnaire (HCQ-14) given to participants before and after a watching a visual probe task used to induce craving.

SECONDARY OUTCOMES:
Secondary Outcome Variable #1a: Cognitive/psychomotor effects (CPT) | +180 minutes post dose
  The cognitive/psychomotor effects of THC and CBD will be assessed using the Continuous Performance Test (CPT). For the CPT, the primary outcome will be the throughput score, which indexes attention/working memory accuracy (i.e. percent of correct responses) and speed (i.e. reaction time).
Secondary Outcome Variable #1b: Cognitive/psychomotor effects (HVLT) | +180 minutes post dose
  The cognitive/psychomotor effects of THC and CBD will be assessed using the Hopkins Verbal Learning Test (HVLT). The primary outcome for the HVLT will be immediate and delayed recall, which index verbal memory.
Secondary Outcome Variable #2a: Abuse potential of combined THC and CBD (MCP) | +480 post dose
  The abuse potential of combined THC and CBD will be assessed using a modified Multiple-Choice Procedure (MCP) at the end of each test session. The primary outcome for the MCP is the crossover point (i.e., the value at which participants choose money over the study medication).
Secondary Outcome Variable #2b: Abuse potential of combined THC and CBD (DEQ) | Up to 8 hours
  The abuse potential of combined THC and CBD will be assessed using the Drug Effects Questionnaire (DEQ) administered at baseline and every 30 minutes. The primary DEQ outcome is the Stimulatory Effects subscale, obtained by averaging participants responses to the items: "Feel High"; "Feel Stimulated"; and "Feel the Drug Strength".
Secondary Outcome Variable #3a: Monitor adverse events from the study medications (SAFTEE) | Baseline ; +480 minutes post dose; One-week after last test session
  To monitor adverse events from the study medications, the Systematic Assessment for Treatment Emergent Events (SAFTEE) will be administered before and after each experimental session and during the one-week follow-up. This is a symptom checklist that has been used successfully in our previous studies to assess possible side effects of study medications. It includes information regarding severity of any presenting side effects, as well as the course of action taken by study staff in response.
Secondary Outcome Variable #3b: Monitor adverse events from the study medications (Cardiovascular) | Up to 8 hours and One-week after last test session
  To monitor cardiovascular effects from the study medications, heart rate and blood pressure will be measured at baseline and every 30 minutes during the experimental sessions, and at the one-week follow-up.

OTHER OUTCOMES:
Central Sensitization | Up to 8 hours
  A central sensitization score will be generated by averaging mechanical temporal summation (TSP), thermal TSP, and conditioned pain modulation (CPM), and after-sensation Z-scores. Negative values will denote antinociception, and positive values will denote pronociception (or central sensitization).
THC and CBD plasma levels | Up to 8 hours
  Whole blood methadone and THC/CBD levels will be obtained to examine potential drug interactions, using liquid chromatography-tandem mass spectrometry (LC-MS/MS). We will determine the peak concentration (Cmax) and time to attain Cmax concentration (Tmax) of each analyte.
Influence of sex | Up to 8 hours
  We will explore if sex moderates the relationships hypothesized in the primary and secondary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Joao P. De Aquino, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper ZD, Haney M. Sex-dependent effects of cannabis-induced analgesia. Drug Alcohol Depend. 2016 Oct 1;167:112-20. doi: 10.1016/j.drugalcdep.2016.08.001. Epub 2016 Aug 5. PMID 27522535
- [Background] Cooper ZD, Craft RM. Sex-Dependent Effects of Cannabis and Cannabinoids: A Translational Perspective. Neuropsychopharmacology. 2018 Jan;43(1):34-51. doi: 10.1038/npp.2017.140. Epub 2017 Jul 17. PMID 28811670
- [Background] Cooper ZD, Haney M. Investigation of sex-dependent effects of cannabis in daily cannabis smokers. Drug Alcohol Depend. 2014 Mar 1;136:85-91. doi: 10.1016/j.drugalcdep.2013.12.013. Epub 2014 Jan 3. PMID 24440051
- [Background] Smith MT Jr, Remeniuk B, Finan PH, Speed TJ, Tompkins DA, Robinson M, Gonzalez K, Bjurstrom MF, Irwin MR. Sex differences in measures of central sensitization and pain sensitivity to experimental sleep disruption: implications for sex differences in chronic pain. Sleep. 2019 Feb 1;42(2):zsy209. doi: 10.1093/sleep/zsy209. PMID 30371854
- [Background] Turri M, Teatini F, Donato F, Zanette G, Tugnoli V, Deotto L, Bonetti B, Squintani G. Pain Modulation after Oromucosal Cannabinoid Spray (SATIVEX(R)) in Patients with Multiple Sclerosis: A Study with Quantitative Sensory Testing and Laser-Evoked Potentials. Medicines (Basel). 2018 Jun 21;5(3):59. doi: 10.3390/medicines5030059. PMID 29933552
- [Background] Dunn KE, Bergeria CL, Huhn AS, Speed TJ, Mun CJ, Vandrey R, Campbell CM. Within-subject, double-blinded, randomized, and placebo-controlled evaluation of the combined effects of the cannabinoid dronabinol and the opioid hydromorphone in a human laboratory pain model. Neuropsychopharmacology. 2021 Jul;46(8):1451-1459. doi: 10.1038/s41386-021-01007-4. Epub 2021 Apr 20. PMID 33879842
- [Background] Matheson J, Mann RE, Sproule B, Huestis MA, Wickens CM, Stoduto G, George TP, Rehm J, Le Foll B, Brands B. Acute and residual mood and cognitive performance of young adults following smoked cannabis. Pharmacol Biochem Behav. 2020 Jul;194:172937. doi: 10.1016/j.pbb.2020.172937. Epub 2020 May 1. PMID 32360692
- [Background] Leweke FM, Rohleder C, Gerth CW, Hellmich M, Pukrop R, Koethe D. Cannabidiol and Amisulpride Improve Cognition in Acute Schizophrenia in an Explorative, Double-Blind, Active-Controlled, Randomized Clinical Trial. Front Pharmacol. 2021 Apr 29;12:614811. doi: 10.3389/fphar.2021.614811. eCollection 2021. PMID 33995015
- [Background] Griffiths RR, Troisi JR, Silverman K, Mumford GK. Multiple-choice procedure: an efficient approach for investigating drug reinforcement in humans. Behav Pharmacol. 1993 Feb;4(1):3-13. PMID 11224166
- [Background] Morean ME, de Wit H, King AC, Sofuoglu M, Rueger SY, O'Malley SS. The drug effects questionnaire: psychometric support across three drug types. Psychopharmacology (Berl). 2013 May;227(1):177-92. doi: 10.1007/s00213-012-2954-z. Epub 2012 Dec 28. PMID 23271193
- [Background] Levine J, Schooler NR. SAFTEE: a technique for the systematic assessment of side effects in clinical trials. Psychopharmacol Bull. 1986;22(2):343-81. No abstract available. PMID 3774930
- [Background] Georgopoulos V, Akin-Akinyosoye K, Zhang W, McWilliams DF, Hendrick P, Walsh DA. Quantitative sensory testing and predicting outcomes for musculoskeletal pain, disability, and negative affect: a systematic review and meta-analysis. Pain. 2019 Sep;160(9):1920-1932. doi: 10.1097/j.pain.0000000000001590. PMID 31045746
- [Background] Yarnitsky D, Granot M, Nahman-Averbuch H, Khamaisi M, Granovsky Y. Conditioned pain modulation predicts duloxetine efficacy in painful diabetic neuropathy. Pain. 2012 Jun;153(6):1193-1198. doi: 10.1016/j.pain.2012.02.021. Epub 2012 Apr 3. PMID 22480803
- [Background] Huestis MA. Human cannabinoid pharmacokinetics. Chem Biodivers. 2007 Aug;4(8):1770-804. doi: 10.1002/cbdv.200790152. No abstract available. PMID 17712819
- [Background] De Aquino JP, Meyerovich J, Xie CZ, Ranganathan M, Compton P, Pittman B, Rogan M, Sofuoglu M. Delta-9-tetrahydrocannabinol modulates pain sensitivity among persons receiving opioid agonist therapy for opioid use disorder: A within-subject, randomized, placebo-controlled laboratory study. Addict Biol. 2023 Sep;28(9):e13317. doi: 10.1111/adb.13317. PMID 37644897
- [Background] De Aquino JP, Bahji A, Gomez O, Sofuoglu M. Alleviation of opioid withdrawal by cannabis and delta-9-tetrahydrocannabinol: A systematic review of observational and experimental human studies. Drug Alcohol Depend. 2022 Dec 1;241:109702. doi: 10.1016/j.drugalcdep.2022.109702. Epub 2022 Nov 18. PMID 36434879
- [Background] Oliveira D, Fontenele R, Weleff J, Sofuoglu M, De Aquino JP. Developing non-opioid therapeutics to alleviate pain among persons with opioid use disorder: a review of the human evidence. Int Rev Psychiatry. 2023 Aug-Sep;35(5-6):377-396. doi: 10.1080/09540261.2023.2229430. Epub 2023 Jun 28. PMID 38299655
- [Background] Costa GPA, Nunes JC, Heringer DL, Anand A, De Aquino JP. The impact of cannabis on non-medical opioid use among individuals receiving pharmacotherapies for opioid use disorder: a systematic review and meta-analysis of longitudinal studies. Am J Drug Alcohol Abuse. 2024 Jan 2;50(1):12-26. doi: 10.1080/00952990.2023.2287406. Epub 2024 Jan 15. PMID 38225727